CLINICAL TRIAL: NCT04002219
Title: Efficacy Evaluation of the Mushroom Beverage on Emotion Regulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Science and Technology Council, Taiwan (Other Government)
Collaborators: National Taiwan University (Other)
Responsible Party: Principal Investigator, Kuan-Pin, Principal Investigator, National Science and Technology Council, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMUH108-REC3-022
Record Dates: First submitted 2019-06-20; First posted 2019-06-28 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Inflammation, Brain; Emotional Problem
MeSH Terms: conditions — Encephalitis

STUDY DESIGN:
Intervention Model Description: A triple-blind, randomized-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active arm (Experimental): Subjects will receive treatment with active beverage containing the active ingredient
  Interventions: Dietary Supplement: beverage containing mushroom-extracts
- Placebo arm (Placebo Comparator): Subjects will receive treatment with placebo beverage not containing the active ingredient
  Interventions: Dietary Supplement: beverage containing mushroom-extracts

INTERVENTIONS:
Dietary Supplement: beverage containing mushroom-extracts — Subjects recruited from both arms will receive treatment and be followed up clinically for 8 weeks.

SUMMARY:
Major Depression Disorder is one of the most common psychiatric disease and has affecting approximately 350 million people in the world. According to World Health Organization's report, it may be the first burden of disease in 2030. Due to the high morbidity and low acceptance in the treatment, it is necessary to find some nature compounds to prevent the disease.

Cordyceps militaris, one of the most treasure Chinese herbs in Asia, contains many kinds of component such as cordycepin, polysaccharide, mannitol. In winter, it appears as an worm in the soil, afterwards, it grows out of the soil and convert into grass in summer. A previous study has demonstrated that Cordyceps militaris has anti-depressive effect in mouse tail suspension test, and in this study we will explore its effect in human subjects.

ELIGIBILITY:
Inclusion Criteria:

1. 21 -items Hamilton Rating Scale for Depression scores 8-17 points upon interview
2. At least 2 weeks not taking antidepressants, antipsychotics or antiepileptics.
3. Understand the whole process of the study and had signed the informed consent form

Exclusion Criteria:

1. Had been diagnosed with severe mental disorder, schizophrenia, bipolar disorder, personality disorder, substance use disorder or alcohol use disorder, or other severe physical illness that is not expected to survive during the intervention period.
2. Currently taking antidepressants or other medication that may impact the study.
3. Expected to be non-adherent.
4. Without sufficient data to confirm safety.
5. Pregnant woman
6. Allergic to fungal products.
7. Currently taking MAO-inhibitors

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Change of subjective depressive symptoms | 8 weeks
  Measured by Beck Depression Inventory-II
Change of objective depressive symptoms | 8 weeks
  Measured by Hamilton Rating Scale for Depression
Change of somatic symptoms | 8 weeks
  Measured by Neurotoxicity Rating Scale, a 39-item self-report scale to evaluate the somatic symptoms such as anorexia, fatigue and pain; higher scores indicate higher severity.
Cortisol level | 8 weeks
  Measured as a stress-related biomarker

CONTACTS AND LOCATIONS:
Overall Officials: Kuan-Pin Su, MD, PhD, Study Director — China Medical University, China
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
The study has not yet fully discuss the plan for IPD opening.